CLINICAL TRIAL: NCT04418141
Title: A Phase I, Open Label, Multi-Center, Dose Escalation Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CN1 in Patients With Advanced Solid Tumors or B-cell Lymphoma
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of CN1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curon Biopharmaceutical (Australia) Co Pty Ltd (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN1-101
Record Dates: First submitted 2020-05-13; First posted 2020-06-05 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumor; B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Five planned CN1 dose levels of 0.03 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg, and 10 mg/kg.
  Subjects will receive CN1 by intravenous infusion (IV) on Day 1 (D1) of each cycle (once every 3 weeks per cycle).
  Interventions: Drug: CN1

INTERVENTIONS:
Drug: CN1 — Participants will receive CN1 by IV infusion on Day 1 of each cycle (every 3 weeks). The 5 planned dose levels are 0.03 mg/kg, 0.3 mg/kg, 1 mg/kg, 3 mg/kg and 10 mg/kg.

SUMMARY:
This study is the first-in-human clinical trial of CN1 to evaluate the safety, tolerability, pharmacokinetic (PK) profile and preliminary efficacy of CN1 in patients with advanced solid tumors or B-cell lymphoma. This study will provide a basis for further clinical development of CN1.

DETAILED DESCRIPTION:
CN1 could promote T cell activation and cytokine secretion, thereby enhancing the function of CD4+ and CD8+ T cells, and could also regulate Treg cells, thus CN1 is considered to enhance the anti-tumor immune response and have potential antitumor activity.

In this multicenter, open-label, dose-escalation Phase I study six dose levels are planned. Participants will receive CN1 by IV infusion on Day 1 of each cycle (every 3 weeks). After completion of treatment cycles, the participant will be assessed by the Principal Investigator and/or Safety Monitoring Committee (SMC).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years old, male or female;
2. Subjects with histologically or cytologically diagnosed advanced malignant solid tumors or B-cell lymphoma who have failed on, or are intolerant to, standard therapy, for whom there are no standard of care regimens, or who are otherwise not eligible for standard therapy at this stage;
3. Subjects with Eastern Cooperative Oncology Group (ECOG) performance score of 0-1;
4. Females must be non-pregnant and non-lactating, and must use an acceptable, highly effective double contraception from screening until the end of the follow-up period.
5. Subjects must be able to understand and sign the paper informed consent before any study specific procedure.

Exclusion Criteria:

1. Received anti-tumor treatment such as radiotherapy, chemotherapy, biotherapy, endocrine therapy, immunotherapy, etc., within 4 weeks prior to the first dose of study drug.
2. Received other investigational agents (not yet approved by any regulatory agency) within 4 weeks prior to the first dose of study drug;
3. Major organ surgery (excluding puncture biopsy) or significant trauma within 4 weeks prior to the first dose of study drug;
4. Systemic application of corticosteroids (prednisone > 10 mg/day or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of study drug;

   * Exceptions: topical, ocular, intra-articular, intranasal, and inhaled corticosteroids, or short-term corticosteroids for prophylaxis (e.g., contrast allergy prophylaxis).
5. Use of live attenuated vaccine within 4 weeks prior to the first dose of study drug;
6. Clinically symptomatic metastases to the central nervous system or meninges, or other evidence of uncontrolled metastases to the central nervous system or meninges of the subject;
7. Active infection and in current need of, or likely to need, intravenous anti-infective therapy;
8. History of immunodeficiency, including history of any positive test result for human immunodeficiency virus (HIV) antibody;
9. Active hepatitis B or hepatitis C virus infection.
10. Subjects with active or previous autoimmune diseases (e.g. systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except subjects with clinically stable autoimmune thyroid disease;
11. Subjects with mental disorders or other conditions that pose high non-compliance risks in the opinion of the investigator;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
To determine dose-limiting toxicity (DLT), maximum tolerated dose (MTD), and/or recommended Phase II dose (RP2D) of CN1 administered to patients with advanced solid tumor or B-cell lymphoma. | 21 Days after the first dose i.e. starting dose level 0.03 mg/kg
  DLT is measured in the observation period of 21 days after the first dose i.e. starting dose level 0.03 mg/kg. if the enrolled subject does not experience a study drug related Grade 2 or higher adverse event (AE) per NCI-Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, the subject will start to receive the next designated dose level of 0.3 mg/kg in the second 21 days dosing cycle.

SECONDARY OUTCOMES:
To assess the safety and tolerability of CN1 in patients with advanced solid tumor or B-cell lymphoma through Physical Exam | From baseline(Week 1) to 90 days after the last dose
  Measured by incidence of abnormal physical examination findings.
To assess the safety and tolerability of CN1 in patients with advanced solid tumor or B-cell lymphoma through Adverse Events/Serious Adverse Events | From baseline(Week 1) to 90 days after the last dose
  Measured by incidence of Adverse Events/Serious Adverse Events. All AEs will be summarized according to the Medical Dictionary for Regulatory Activities (MedDRA) v23.0 or higher and the severity will be categorized by CTCAE v5.0. The summary of all AEs will be focused on the treatment-emergent adverse events (TEAEs). A TEAE is defined as any AE that starts after the first dose of study drug till 90 +/- 7 days after the last dose of study drug.
To assess the pharmacokinetic (PK) profile of CN1 in patients with advanced solid tumor or B-cell lymphoma through Area under the plasma concentration-time curve | Measurement is through treatment completion starting from Week 1 up to End of Treatment, assessed up to an average of 10 weeks.
  The following parameter is used for evaluation during PK assessments: Area under the plasma concentration-time curve (AUC0-t, AUC0- ∞, AUC0-τ)
To assess the pharmacokinetic (PK) profile of CN1 in patients with advanced solid tumor or B-cell lymphoma through Tmax | Measurement is through treatment completion starting from Week 1 up to End of Treatment, assessed up to an average of 10 weeks.
  The following parameter is used for evaluation during PK assessments: Time to maximum (Tmax)
To assess the pharmacokinetic (PK) profile of CN1 in patients with advanced solid tumor or B-cell lymphoma through Apparent volume of distribution at steady state | Measurement is through treatment completion starting from Week 1 up to End of Treatment, assessed up to an average of 10 weeks.
  The following parameter is used for evaluation during PK assessments: Apparent volume of distribution at steady state (Vss)
To assess the pharmacokinetic (PK) profile of CN1 in patients with advanced solid tumor or B-cell lymphoma through Accumulation factor based on AUC 0-τ | Measurement is through treatment completion starting from Week 1 up to End of Treatment, assessed up to an average of 10 weeks.
  The following parameter is used for evaluation during PK assessments: Accumulation factor based on AUC 0-τ (R AUC0-τ)
To assess the immunogenicity to CN1 in patients with advanced solid tumor or B-cell lymphoma through ADA testing | Measurement is through treatment completion starting from Week 1 up to End of Treatment, assessed up to an average of 10 weeks.
  A validated analysis method will be used for detection of anti-drug antibodies (ADA).
To explore the anti-tumor efficacy of CN1 in patients with advanced solid tumor or B-cell lymphoma through ORR analysis | Measurement is from Week 1, until the 90 days after the last dose, date of first documented progression or unacceptable toxicity, withdrawal of consent, subject being lost to follow-up, or death, whichever occurs first.
  Assessed by the number of participants with objective response (ORR)
To explore the anti-tumor efficacy of CN1 in patients with advanced solid tumor or B-cell lymphoma through DCR analysis. | Measurement is from Week 1, until the 90 days after the last dose, date of first documented progression or unacceptable toxicity, withdrawal of consent, subject being lost to follow-up, or death, whichever occurs first.
  Assessed by the number of participants with Disease Control (DCR)
To explore the anti-tumor efficacy of CN1 in patients with advanced solid tumor or B-cell lymphoma through DoR analysis. | Measurement is from Week 1, until the 90 days after the last dose, date of first documented progression or unacceptable toxicity, withdrawal of consent, subject being lost to follow-up, or death, whichever occurs first.
  Assessed by the number of participants with Duration of Response (DoR)

CONTACTS AND LOCATIONS:
Overall Officials: John Park, Principal Investigator — Macquarie University Hospital; Jim Coward, Principal Investigator — Icon Cancer Centre (Brisbane); Daniel Brungs, Principal Investigator — Illawarra Cancer Care Centre (Wollongong); Gary Richardson, Principal Investigator — Cabrini Hospital (Melbourne)
Locations (1):
- Mater Medical Centre, Brisbane, Queensland, Austria

IPD SHARING:
Plan to Share IPD: No